CLINICAL TRIAL: NCT05615168
Title: Use of Hypotension Prediction Index to Reduce Intraoperative Hypotension in Major Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Andrej Šribar, Prinicipal investigator, Head of division of cardiovascular anesthesiology, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022/1807-03
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hypotension During Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AcumenIQ - HPI guided hemodynamic optimization (Experimental): HPI guided hypotension prediction alarms... Interventions based on SVV (fluid), dp/dt (inotropes), EAdyn (pressors)
  Interventions: Diagnostic Test: "Acumen IQ" guided hemodynamic optimization
- Flotrac - conventional GDT guided hemodynamic optimization (Active Comparator): GDT guided hemodynamic optimization - MAP > 65 mmHg, CI ≥ 2.4 l/min/m2, SVI ≥ 30 ml/beat/m2 and SVRI 1700-2400 dyn·s·cm-5/m2
  Interventions: Diagnostic Test: "Flotrac" guided hemodynamic optimization

INTERVENTIONS:
Diagnostic Test: "Acumen IQ" guided hemodynamic optimization — Hypotension prediction index (HPI) available with the Edwards "Acumen IQ" sensor will be used as an early warning system and a "diagnostic screen" will be used to guide therapeutic interventions.
  Arms: AcumenIQ - HPI guided hemodynamic optimization
Diagnostic Test: "Flotrac" guided hemodynamic optimization — Therapeutic interventions guided by real time monitored hemodynamic parameters as measured by Edwards "Flotrac" sensor.
  Arms: Flotrac - conventional GDT guided hemodynamic optimization

SUMMARY:
Intraoperative hypotension is linked to increased incidence of perioperative adverse events such as myocardial and cerebrovascular infarction and acute kidney injury. Hypotension prediction index (HPI) is a novel machine learning guided algorithm which can predict hypotensive events using high fidelity analysis of pulse-wave contour. Goal of this trial is to determine whether use of HPI can reduce the number and duration of hypotensive events in patients undergoing major thoracic procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* patients scheduled for elective major thoracic procedure (lung resection, pleurectomy or resection of the esophagus)
* planned thoracotomy and intraoperative period of one lung ventilation
* planned postoperative admission to the ICU

Exclusion criteria:

* persistent atrial fibrillation
* structural heart defects (shunting or moderate to severe valvular anomalies)
* preoperative serum hemoglobin levels < 120 g/L
* severe heart failure classified as New York Heart Association (NYHA) grade IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Time weighted average of area under hypotensive threshold | During surgery

SECONDARY OUTCOMES:
Cumulative duration of hypotension | During surgery
Number of hypotensive events | During surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
Will share anonymized data after article publication